CLINICAL TRIAL: NCT04471896
Title: Examining the Impact of Infrared Light Therapy Device on Cosmetic Skin Health
Brief Title: Joovvin' for Your Skin Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProofPilot (Industry)
Collaborators: Joovv (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2521
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Skin Inflammation; Acne; Skin Diseases; Dermatological Non-Disease; Skin Condition; Eczema
MeSH Terms: conditions — Dermatitis; Acne Vulgaris; Skin Diseases; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Participants will receive an infrared therapy device for use at home for 60 days. Participants will use the device every day for 10-20 minutes during the intervention period.
  Interventions: Device: Joovv Mini

INTERVENTIONS:
Device: Joovv Mini — Infrared light therapy uses certain wavelengths of light that are delivered to the face. This study will use the Joovv Mini.
  Other Names: Infrared light therapy device

SUMMARY:
Sixty day single arm trial examining self-report and remote dermatology assessment of cosmetic skin health after daily 10-20 minute sessions with an infrared light therapy device (the Joovv Mini)

ELIGIBILITY:
Inclusion Criteria:

* willingness to use device for 60 days
* willingness to place security deposit on device of $149.99
* US resident with an address than can accept UPS deliveries
* 18 years old
* no serious medical conditions
* no medically treatable skin diseases
* willingness to take a selfie with mobile phone

Exclusion Criteria:

* Retinoid use
* prior use of light therapy within the past 6 months
* pregnant or nursing
* dietary supplements for skin, hair or nail health

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Blinded Dermatology Assessment of Facial Skin Health | 60 day
  Comparison over timepoints of physician assessment of facial features at rest and smile to the Glogau & custom wrinkle selfie scale
Changes in Self-Report Skin, Hair & Nail Health and Satisfaction | 60 day
  A custom self report survey on cosmetic skin health satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot (Virtual Study: https://p.proofpilot.com), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided